CLINICAL TRIAL: NCT03941080
Title: Gut Microbiome Dynamics in Metastasized or Irresectable Colorectal Cancer: Initiating a Prospective Multicenter Cohort (GIMICC)
Brief Title: Gut Microbiome Dynamics in Metastasized or Irresectable Colorectal Cancer
Acronym: GIMICC
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 201900296
Record Dates: First submitted 2019-04-29; First posted 2019-05-07 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer Metastatic
Keywords: colorectal cancer; gut microbiome
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal sample and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GIMICC: Adult patients with newly diagnosed metastasized or irresectable CRC with an indication for standard palliative systemic anti-tumor treatment.
  Interventions: Diagnostic Test: fecal sample; Behavioral: questionnaire; Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: fecal sample — patients will collect fecal samples at home prior to treatment and at 3 months after start of treatment at the time of response evaluation using a standard stool-collection-kit.
Behavioral: questionnaire — At the day of stool sampling, patients fill out a brief questionnaire about established factors that can change the microbiome such concurrent use of antibiotics and proton pump inhibitors.
Diagnostic Test: Blood sample — 4 tubes of blood are collected prior to treatment and at 3 months after start of treatment at the time of response evaluation and sent to the UMCG for storage.

SUMMARY:
In this study the characteristics and alterations of the gut microbiome during chemotherapy for metastasized or irresectable CRC are studied, as well as the relation between the gut microbiome and the effects of chemotherapy.

DETAILED DESCRIPTION:
Although systemic treatment for metastasized or irresectable colorectal cancer (CRC) is becoming increasingly effective, overall survival is still poor and side effects of current treatment modalities are substantial. There is an urgent need for novel therapies, and in addition, better predictive tools are needed to select the right drug to the right patient. New data suggest that modulation of the microbiome of the gut might provide opportunities to increase anti-tumor efficacy of immunotherapy. Whereas the relation between the gut microbiome and immunotherapy is intensively studied, the relation between the gut microbiome and efficacy of conventional chemotherapy is unknown. A better understanding of the composition, function and dynamics of the gut microbiome before and during chemotherapy might help to identify factors that can be influenced during the treatment of patients with metastasized or irresectable CRC.

Therefore, in this study the characteristics and alterations of the gut microbiome during chemotherapy for metastasized or irresectable CRC are studied, as well as the relation between the gut microbiome and the effects of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with histologically confirmed CRC with an indication for palliative systemic anti-tumor therapy (ANY combination of chemotherapy with/without anti-VEGF of anti-EGFR therapy)
* Measurable disease according to RECIST v1.1.
* Stored pathological specimens available
* Life expectancy ≥ 12 weeks
* Signed Informed Consent Form
* Ability to comply with protocol

Exclusion Criteria:

* Previous (neo)adjuvant chemotherapy < 6 months
* Previous radiotherapy on the small or large intestine < 1month
* Previous surgery of the small or large intestine < 1 month
* Uncontrolled inflammatory bowel disease
* Participation in a study with a potential effect on the gut microbiome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present in the hospitals of the North Netherlands Colorectal Cancer Network. The participating hospitals together cover 10% of the Dutch population. Given that 13.000 patients yearly are diagnosed with colorectal cancer of which one third will develop metastatic or irresectable disease (www.iknl.nl), in the hospitals participating in this study 400 potential patients will present. Taking into account that about 50% do not fulfil in- and exclusion criteria or will refuse to participate, about 200 patients per year are expected to be included.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Prediction of response to conventional systemic anti-tumor therapy conventional systemic anti-tumor therapy for metastatic or irresectable colorectal cancer | 2 years
  To determine which bacteria species in the microbiome predict response to conventional systemic anti-tumor therapy according to RECIST v1.1 for metastatic or irresectable colorectal cancer

SECONDARY OUTCOMES:
Prediction of serious side effects to conventional systemic anti-tumor therapy for metastatic or irresectable colorectal cancer | 2 years
  To determine which bacteria strains in the microbiome predict serious side effects (grade 3/4 according to CTCAE v4.03) to conventional systemic anti-tumor therapy for metastatic or irresectable colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: J. J. de Haan, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (10):
- Netherlands (10):
  - Wilhelmina Ziekenhuis, Assen
  - Ziekenhuis Nij Smellinghe, Drachten
  - Treant Zorggroep, Emmen
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Martini Ziekenhuis, Groningen
  - Tjongerschans Ziekenhuis, Heerenveen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Ommelander Ziekenhuis Groep, Scheemda
  - Antonius Zorggroep, Sneek